CLINICAL TRIAL: NCT00858754
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of Subcutaneous Methylnaltrexone for the Treatment of Opioid-Induced Constipation in Subjects With Cancer-Related Pain
Brief Title: Study Evaluating Safety & Efficacy of Subcutaneous Methylnaltrexone on Opioid-Induced Constipation in Cancer Subjects
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn [This study was terminated early by Wyeth, prior to dosing any subjects, for business reasons not related to safety.
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200K1-4006
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Opioid-Induced Constipation
Keywords: opioid induced constipation; Cancer patients; methylnaltrexone
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Active Drug (Experimental): Methylnaltrexone
  Interventions: Drug: methylnaltrexone
- Group 2 Non-Active Drug (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylnaltrexone
  Other Names: MOA-728
  Arms: Group 1 Active Drug
Drug: placebo
  Other Names: Inactive
  Arms: Group 2 Non-Active Drug

SUMMARY:
This purpose of this study is to evaluate the safety and effectiveness of a subcutaneous (injection beneath the skin) form of methylnaltrexone in subjects who have cancer-related pain and constipation from taking opioids. The length of participation will be up to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is a man or woman aged 18 years or older.
* Has a body weight >= 38 kg.
* Has cancer (active or in remission), and has cancer-related pain (ie, pain due to cancer or treatment of cancer).
* Has a life expectancy of >= 6 months.
* Has a performance status of 0, 1, or 2 based on the Eastern Cooperative Oncology Group (ECOG) scale.
* Is taking opioids for cancer-related pain, and not just as-needed doses.
* Has a diagnosis of OIC as determined by the investigator.
* Is willing to follow the protocol instructions on laxative use during the study.

Exclusion Criteria:

* Has a history of chronic constipation before starting opioids.
* Has renal disease receiving dialysis.
* Has an ostomy for stools.
* Is a pregnant or breastfeeding woman.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Bowel movement within 4 hours after the first dose. Collection of adverse events, vital signs measurements, and laboratory assessments. | 1 Day

SECONDARY OUTCOMES:
1. Bowel movements within 4 hours after at least 2 of the first 4 doses. 2. Bowel movements within 4 hours after all doses. 3. The time to bowel movement after the first dose. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (8):
- United States (4):
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Lancaster, California
  - Pfizer Investigational Site, Flat Rock, North Carolina
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Edmonton, Alberta, Canada
- Pfizer Investigational Site, Villejuif, France
- Pfizer Investigational Site, El Palmar, Murcia/Spain, Spain
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3200K1-4006&StudyName=Study%20Evaluating%20Safety%20%26%20Efficacy%20of%20Subcutaneous%20Methylnaltrexone%20on%20Opioid-Induced%20Constipation%20in%20Cancer%20Subjects